CLINICAL TRIAL: NCT00761111
Title: Could a Simple Information Booklet Modify Low Back Pain Patients Beliefs After Lumbar Discectomy?
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Pascale GIVRON, CHU Clermont-Ferrand
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: CHU63-0023
Record Dates: First submitted 2007-08-22; First posted 2008-09-29 (Estimated); Last update posted 2008-10-08 (Estimated); Status verified 2008-10

CONDITIONS: Back Pain
Keywords: information booklet; low back beliefs; education; disc hernia; discectomy; A common monoradicular sciatica; on a slipped disc; with a clinical radio; agreement requiring a surgical treatment; carried out; one duration; of evolution higher; than four weeks; at naive subjects; of any rachidian interventional treatment; after failure of an good ambulatory
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Behavioral: Assessment of the Your Back Operation — to translate and assess an evidence based educational booklet on low back pain patients beliefs after lumbar discectomy

SUMMARY:
The purpose of this study is to translate and assess an evidence based educational booklet on low back pain patients beliefs after lumbar discectomy.

DETAILED DESCRIPTION:
A translation / back-translation of the Your back operation was performed and a before / after prospective study was realized. Main outcome assessment was the Quebec Questionnaire. Demographic data, personal medical sciatica pain history, graduation of the whole subject were recorded. Acceptability of the booklet was also measured.

ELIGIBILITY:
Inclusion Criteria:

* A common monoradicular sciatica on a slipped disc with a clinical radio agreement requiring a surgical treatment, after failure of an good ambulatory treatment carried out, one duration of evolution higher than four weeks at naive subjects of any rachidian intervention

Exclusion Criteria:

* People presenting a cruralgia, a secondary sciatica (epiduritis, osseous metastasis...) or without relationship with a slipped disc (spinal stenosis), an lesion biradicular, an horse tail syndrome, an important motor deficit (muscular testing < 3)
* Cognitive, auditive, major visual disorders or any subject which does not have a good comprehension of spoken French and/or writing, or having recourse to a third for reading and supplementing a document
* Subjects presenting a peripheral neuropathy, a severe and evolved diabetes, a cardiac insufficiency, dialysed subject
* People observing a treatment which included psychotropics for more than three months (other that light hypnotic) because of the disturbances of vigilance and memory

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2007-06; Primary Completion 2008-05 (Estimated)

PRIMARY OUTCOMES:
Quebec Questionnaire | after lumbar discectomy

SECONDARY OUTCOMES:
FABQ Questionnaire | after lumbar discectomy
Rachidian and radicular painful intensity | after lumbar discectomy

CONTACTS AND LOCATIONS:
Overall Officials: Givron Pascale, Dr, Principal Investigator

REFERENCES:
- [Derived] Claus D, Coudeyre E, Chazal J, Irthum B, Mulliez A, Givron P. An evidence-based information booklet helps reduce fear-avoidance beliefs after first-time discectomy for disc prolapse. Ann Phys Rehabil Med. 2017 Apr;60(2):68-73. doi: 10.1016/j.rehab.2015.10.008. Epub 2016 Jan 6. PMID 26776321